CLINICAL TRIAL: NCT02115412
Title: Validation of Medication Non-adherence Model (UK)
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: PhilipsResearch-2007-0116
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus; Chronic Obstructive Pulmonary Disease; Chronic Illness; Primary Care; Medication Management at Home
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- medication non-adherence

SUMMARY:
Research has shown that nearly 50% of patients with chronic conditions around the globe do not adhere to their prescribed medicine, leading to enormous cost to the healthcare providers. Non-adherence can be due to various forms and have multiple causes.

To address this need, Philips Research has developed Medication Non-adherence model. This tool will help in developing a systemic way of assessing medication non-adherence and providing decision support for targeted intervention to healthcare professionals. The aim of this study is to validate this model with 750 chronically ill patients in UK.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic disease between 18 -89 years old.
* Chronic medication use (> 3 medications; excluding analgesic, ointment and eye drop medication)
* Patients registered with a given Pharmacy at least 1 year before entering into the study.

Exclusion Criteria:

* Patients who are illiterate in English.
* Patients who are unable to give consent to the study.
* Enrolled in another clinical trial, which requires change in their routinely medication.
* Patients currently using automatic medication reminder services (excluding the pharmacy service).
* Patients with dementia or any other mental conditions, that might affects the accuracy of the answers provided.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic illness taking more than 3 medications. These patients will be between the age of 18 - 89
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adherence determinants | 6 months
  Self-reported behavioral questionnaire completed at 3 monthly intervals

SECONDARY OUTCOMES:
Medication usage | 18 months
  Collecting refill data from the pharmacy where patients are registered to. Time Frame: 18 months (12 month prior to enrollment + 6 months during the study

OTHER OUTCOMES:
Adverse Events | 18 months
  Any adverse events (eg: hospitalisation, elective surgeries), which may have resulted change in their daily medication routine Time Frame: 18 months, meaning 12 month prior to enrollment + 6 months during the study

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Swan Lane Medical Centre, Bolton, Greater Manchester
  - Vida Health, 39 Gayton Road, Kings Lynn, Norfolk
  - Rosedale Surgery, Carlton Colville, Lowestoft, Suffolk
  - Wymondham Medical Practice, Norfolk